CLINICAL TRIAL: NCT05636033
Title: Semantic Networks in Alcohol Use Disorder Patients: Exploratory Study
Acronym: ALCOOLNET
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C22-01; 2022-A01903-40 (Registry Identifier: ID RCB)
Record Dates: First submitted 2022-11-03; First posted 2022-12-05 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Use Disorder
Keywords: alcohol use disorder; semantic association; semantic networks; cognition
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Alcohol use disorder patients
- Healthy controls

SUMMARY:
Alcohol Use Disorder (AUD) is a major public health problem, characterized by a high rate of relapse. Chronic and excessive alcohol consumption notably induces frontal brain alterations and cognitive impairments such as executive dysfunction and an attentional bias for alcohol, participating to the risk of relapse. In effect, AUD patients preferentially process alcohol-related cues, which could reflect a reorganization of the patients' semantic network. The investigators hypothesize that in AUD patients, semantic associations in memory are reorganized with a higher centrality of alcohol-related elements. To the investigators knowledge, no studies have explored semantic associations and/or semantic networks in AUD.

A study, conducted in patients with neurological damage, showed that frontal lesions are associated with excessive strength in semantic associations, and difficulties to generate remote associations. This excessive strength in semantic associations could reduce the ability to inhibit automatisms and to adapt to new context.

Objective: The objective of this study is to explore whether and how AUD patients have a different organization of semantic associations than healthy controls, and whether this reorganization influences the alcohol consumption over the months following the withdrawal. The investigators will also explore how it relates to neuropsychological assessment of flexibility, executive functions, and impulsivity. To these purposes, the investigators will use two original verbal tasks (Free Generation of Associates Task, FGAT and Associative Judgment Task, AJT) assessing word associations and allowing the estimation of semantic networks using graph theory, in combination with neuropsychological testing, in AUD patients and in healthy controls.

Methods: This study will include a group of 30 AUD patients and a group of 30 healthy controls. Both groups will be assessed twice, at baseline (T1; early in abstinence for AUD patients) and after a three-month period (T3). For the two groups, T1 and T3 assessments will include the two semantic association tasks (FGAT and AJT). For AUD patients, assessments will also involve neuropsychological testing of impulsivity, flexibility, and attentional bias. Besides, in AUD patients, data about alcohol consumptions will be collected six weeks (T2) and three months (T3) following the baseline assessment to classify patients as relapsers or abstainers.

ELIGIBILITY:
Inclusion Criteria:

For alcohol use disorder patients

* Severe alcohol use disorder
* French as mother tongue
* Right-hander
* Patient abstinent from alcohol since 15 to 30 days at the inclusion
* Patient free from benzodiazepine since at least 48hours at the inclusion
* Patient who gave his informed written consent
* Currently in outpatient or inpatient care

For healthy controls

* French as mother tongue
* Right-hander
* Participant who gave his informed written consent

Exclusion Criteria:

For alcohol use disorder patients

* Patient under guardianship or under justice safeguard measures
* Patient under measure of therapeutic injunction
* Pregnancy or breastfeeding declared
* Meeting Diagnostic and Statistical Manual 5 (DSM) criteria for substance use disorder other than Tobacco
* Meeting DSM-5 criteria for non substance use disorder
* Patient presenting severe or progressive disease that interfere with experimental tasks, such as neurological diseases (TBI, epilepsy, stoke) , hepatic diseases, cancer, HIV, Hepatitis C Virus (HCV), and unstable psychiatric comorbidities.

For healthy controls

* Participant under guardianship or under justice safeguard measures
* Participant under measure of therapeutic injunction
* Pregnancy or breastfeeding declared
* Meeting DSM-5 criteria for alcohol use disorder
* Meeting DSM-5 criteria for substance use disorder other than Tobacco
* Meeting DSM-5 criteria for non substance use disorder
* Currently under benzodiazepine
* Participant presenting severe or progressive disease that interfere with experimental tasks, such as neurological diseases (TBI, epilepsy, stoke) , hepatic diseases, cancer, HIV, HCV, and unstable psychiatric comorbidities.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Two groups of participants will be included in this study. The first one consists of a pool of alcohol use disorder, the second one consists of a pool of healthy controls ; they will be matched as much as possible on age, gender, and educational level.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Description of the semantic associations using FGAT | At baseline (T1)
  The Free Generation Associated Tasks will be used in Alcohol use disorder patients and Healthy controls
Description of the semantic associations using AJT | At baseline (T1)
  The Associative Judgment Task will be used in Alcohol use disorder patients and Healthy controls

SECONDARY OUTCOMES:
Impact of medications on the semantic association performance | At baseline (T1)
Impact of age on the semantic association performance | At baseline (T1)
Impact of the study level on the semantic association performance | At baseline (T1)
Impact of gender on the semantic association performance | At baseline (T1)
Impact of the duration of dependence on the semantic association performance | At baseline (T1)
Impact of cognitive performance on the semantic association performance | At baseline (T1)
  The Go /No Go performance will be collected in Alcohol use disorder patients
Test of the predictive value of FGAT performance assessed at T1 on alcohol consumption during the six weeks following the Baseline | Baseline (T1) for FGAT ; T2 (6 weeks after T1) for alcohol consumption
Test of the predictive value of AJT performance assessed at T1 on alcohol consumption during the six weeks following the Baseline | Baseline (T1) for AJT ; T2 (6 weeks after T1) for alcohol consumption
Test of the predictive value of FGAT performance assessed at T1 on alcohol consumption during the three months following the Baseline | Baseline (T1) for FGAT ; T3 (3 months after T1) for alcohol consumption
Test of the predictive value of AJT performance assessed at T1 on alcohol consumption during the three months following the Baseline | Baseline (T1) for AJT ; T3 (3 months after T1) for alcohol consumption
Evolution of FGAT performance, comparison between alcohol use disorder patients and healthy controls | T1 (baseline) and T3 (3 months after baseline)
Evolution of AJT performance, comparison between alcohol use disorder patients and healthy controls | T1 (baseline) and T3 (3 months after baseline)
Link between the evolution of FGAT performance and the level of alcohol consumption | Baseline (T1) for FGAT and 3 months after baseline (T3) for FGAT and the level of alcohol consumption)
  The level of alcohol consumption will be assessed using the Timeline Followback method
Link between the evolution of AJT performance and alcohol consumption | Baseline (T1) for AJT and 3 months after baseline (T3) for AJT and the level of alcohol consumption)
  The level of alcohol consumption will be assessed using the Timeline Followback method
Link between the evolution of FGAT performance and the evolution of cognitive performance | Baseline (T1) and 3 months after baseline (T3)
  The Go /No Go performance will be used in alcohol use disorder patients
Link between the evolution of AJT performance and the evolution of cognitive performance | Baseline (T1) and 3 months after baseline (T3)
  The Go /No Go performance will be used in alcohol use disorder patients

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Dereux, PH (MD), Principal Investigator — APHP
Locations (1):
- Fernand Widal Hospital, Paris, Île-de-France Region, France